CLINICAL TRIAL: NCT00894114
Title: A Probe Study of the Safety, Tolerability, and Immunogenicity of a 1-Dose Regimen of the MRKAd5 HIV-1 Gag Vaccine Versus the ALVAC-HIV (vCP205) Vaccine in Healthy Adults Who Previously Received a 3-Dose Regimen of MRKAd5, Ad5, or Placebo in Merck V520 Protocols 007 or 012
Brief Title: A Study of Safety, Tolerability and Immunogenicity of a 1-Dose Regimen of MRKAd5 HIV-1 Gag Vaccine Versus the ALVAC_HIV Vaccine (V520-019)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V520-019; 2009_585
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Stratum 1 (Other): Placebo recipients in the parent protocol (Merck V520 Protocols 007 or 012) will receive ALVAC-HIV Vaccine
  Interventions: Biological: Comparator: ALVAC-HIV vaccine
- Stratum 2 (Experimental): Nonresponders who received active vaccine in parent protocol will be randomized to receive ALVAC-HIV vaccine or MRKAd5 HIV-1 gag vaccine
  Interventions: Biological: V520; Biological: Comparator: ALVAC-HIV vaccine
- Stratum 3 (Experimental): Low responders who received active vaccine in the parent protocol will be randomized to receive ALVAC-HIV vaccine or MRKAd5 HIV-1 gag vaccine
  Interventions: Biological: V520; Biological: Comparator: ALVAC-HIV vaccine
- Stratum 4 (Experimental): High responders who received active vaccine in the parent protocol will be randomized to receive ALVAC-HIV vaccine or MRKAd5 HIV-1 gag vaccine
  Interventions: Biological: V520; Biological: Comparator: ALVAC-HIV vaccine

INTERVENTIONS:
Biological: V520 — MRKAd5 HIV-1 gag vaccine, a single dose 1.0 mL intramuscular injection
  Arms: Stratum 2; Stratum 3; Stratum 4
Biological: Comparator: ALVAC-HIV vaccine — A single dose 0.1 intramuscular injection

SUMMARY:
This study is designed to determine whether patients previously primed with Ad5 of MRKAd5 HIV-1 gag vaccine respond better when boosted with ALVAC-HIV vaccine than when boosted with MKRAd5 HIV-1 gag vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously enrolled in Merck HIV Vaccine study V520 Protocol 007 or 012, and received the complete 3-dose regimen during participation
* Subject is in good general health
* Subject is not infected with HIV
* Subject agrees not to donate blood during the first 52 weeks of the study
* Subject agrees not to donate sperm during the first 12 weeks of the study
* Subject who is of reproductive potential agrees to use an acceptable method of birth control through Week 12 of the study

Exclusion Criteria:

* Subject has been administered immune globulin or blood product 3 months prior to receiving study vaccination
* Subject has been vaccinated with a live virus vaccine in the past 30 days
* Subject has been vaccinated with an inactivated vaccine in the past 14 days
* Subject has an active medical disease
* Subject is taking daily required prescription drugs
* Female subject is pregnant, breastfeeding or expecting to conceive
* Subject is positive for HIV
* Subject has used injection drug within the past year
* Subject has a sexual partner that is infected with HIV
* Subject has a sexual partner that is an active injection drug user
* Subject has been treated for or diagnosed with a new sexually transmitted disease in the past 6 months
* Subject engaged in unprotected intercourse with more than 2 persons in the previous 6 months
* Subject engaged in protected intercourse with more than 4 persons in the previous 6 months
* Subject has previously participated in an HIV vaccine clinical trial (other than Merck V520 Protocols 007 and 012)
* Subject weighs less than 110 lbs.
* Subject has a recent history of alcohol abuse
* Subject intends to donate blood in the first 52 weeks of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ALVAC-HIV or MRKAd5 HIV-1 vaccine in subjects who previously received a 3-dose regimen of Ad5 HIV-1 gag vaccine measured by number of injection-site adverse experiences (AE), non serious systemic AE, lab AE, serious AE. | Injection-site AE up to 5 days after vaccination, non-serious systemic AE and Lab AE up to 29 days after vaccination, serious AE for the entire study period (Week 260).

SECONDARY OUTCOMES:
immunogenicity of a single-dose regimen of the ALVAC-HIV vaccine or MRKAd5 HIV-1 vaccine measured by various assays | 4 weeks following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC